CLINICAL TRIAL: NCT02639910
Title: A Phase II, Two-Cohort, Open-Label, Multicenter Study to Evaluate the Safety and Preliminary Efficacy of MOR00208 Combined With Idelalisib or Venetoclax in Patients With Relapsed or Refractory CLL/SLL Previously Treated With Bruton's Tyrosine Kinase (BTK) Inhibitor
Brief Title: Study to Evaluate Safety and Preliminary Efficacy of Tafasitamab With Idelalisib or Venetoclax in R/R CLL/SLL Patients Pretreated With BTKi
Acronym: COSMOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR208C205
Record Dates: First submitted 2015-12-15; First posted 2015-12-28 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CD19; MOR208; MOR00208; CLL; SLL; COSMOS; tafasitamab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tafasitamab; idelalisib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (Experimental): tafasitamab (MOR208) in combination with idelalisib
  Interventions: Biological: Tafasitamab; Drug: Idelalisib
- Cohort B (Experimental): tafasitamab (MOR208) in combination with venetoclax
  Interventions: Biological: Tafasitamab; Drug: Venetoclax

INTERVENTIONS:
Biological: Tafasitamab — tafasitamab (MOR208) dose: 12 mg/kg intravenous infusion
  Other Names: MOR208; MOR00208
Drug: Idelalisib — idelalisib dose: 150 mg twice daily orally
  Other Names: Zydelig; GS-1101 or CAL-101
  Arms: Cohort A
Drug: Venetoclax — venetoclax dose: 400 mg once daily orally
  Other Names: Venclexta, Venclyxto; ABT-199
  Arms: Cohort B

SUMMARY:
This is a two-cohort, multicenter, open-label study of tafasitamab (MOR208) combined with idelalisib or venetoclax in adult patients with R/R CLL or R/R SLL pretreated with a BTK inhibitor (e.g., ibrutinib) as single agent or as part of combination therapy. Patients completing the study treatment are invited to participate in an optional biomarker sub-study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical safety and preliminary efficacy of tafasitamab (MOR208) combined with idelalisib or venetoclax. The study will include safety run-in phase for each cohort with an evaluation of the safety data by an Independent Data Monitoring Committee.

An optional sub-study has been introduced to collect biological samples for investigations on biomarkers (e.g., CD19 expression) after tafasitamab treatment.

ELIGIBILITY:
Major inclusion criteria

Diagnosis/Trial Population

* Chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL):

  * history of diagnosis of CLL or SLL that meets IWCLL diagnostic criteria
  * histologically confirmed diagnosis of SLL by lymph node biopsy
  * indication for treatment as defined by the IWCLL guidelines
* Patients must have both of the following:

  * relapsed or refractory disease while receiving a BTKi therapy or intolerance of such therapy
  * single-agent or combination therapy with a BTKi for at least one month must be the patient's most recent prior anticancer therapy
* ECOG performance status of 0 to 2
* Patients with a past medical history of autologous or allogeneic stem cell transplantation must exhibit full hematological recovery

Laboratory Values

• Patients must meet adequate bone marrow function and adequate hepatic and renal function

Other Inclusion Criteria

• Females of childbearing potential must use a highly effective method of contraception

Major exclusion criteria

Diagnosis

• Patients who have:

* non-Hodgkin's lymphomas other than CLL/SLL
* transformed CLL/SLL or Richter's syndrome
* active and uncontrolled autoimmune cytopenia

Previous and Current Treatment

* Patients who have received treatment with a BTK inhibitor within 5 days prior to Day 1 dosing
* Patients who have, within 14 days prior to D1 dosing:

  * not discontinued CD20-targeted therapy, chemotherapy, radiotherapy, investigational anticancer therapy or other lymphoma specific therapy
  * systemic corticosteroids in doses greater than prednisone equivalent to 20 mg/day with the exception of patients with signs of rapidly progressing disease
  * received live vaccines with the exception of vaccination against influenza with inactivated virus or for pneumococcal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anke Muth, Study Director — Clinical Development, MorphoSys AG
Locations (17):
- United States (3):
  - Clinical Study Site, Jacksonville, Florida
  - Clinical Study Site, Rochester, Minnesota
  - Clinical Study Site, Columbus, Ohio
- Austria (3):
  - Clinical Study Site, Graz
  - Clinical Study Site, Salzburg
  - Clinical Study Site, Vienna
- Germany (3):
  - Clinical Study Site, Dresden
  - Clinical Study Site, Leipzig
  - Clinical Study Site, München
- Italy (2):
  - Clinical Study Site, Brescia
  - Clinical Study Site, Milan
- Poland (4):
  - Clinical Study Site, Gdansk
  - Clinical Study Site, Krakow
  - Clinical Study Site, Lublin
  - Clinical Study Site, Opole
- United Kingdom (2):
  - Clinical Study Site, Bournemouth
  - Clinical Study Site, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staber PB, Jurczak W, Greil R, Vucinic V, Middeke JM, Montillo M, Munir T, Neumeister P, Schetelig J, Stilgenbauer S, Striebel F, Dirnberger-Hertweck M, Weirather J, Brugger W, Kelemen P, Wendtner CM, Woyach JA. Tafasitamab combined with idelalisib or venetoclax in patients with CLL previously treated with a BTK inhibitor. Leuk Lymphoma. 2021 Dec;62(14):3440-3451. doi: 10.1080/10428194.2021.1964020. Epub 2021 Aug 20. PMID 34414843

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Tafasitamab+Idelalisib): Tafasitamab (MOR208) in combination with idelalisib
  Tafasitamab dose: 12 mg/kg intravenous infusion
  Idelalisib dose: 150 mg twice daily orally
- Cohort B (Tafasitamab+Venetoclax): Tafasitamab (MOR208) in combination with venetoclax
  Tafasitamab dose: 12 mg/kg intravenous infusion
  Venetoclax dose: 400 mg once daily orally
Period: Overall Study
Arm/Group | Cohort A (Tafasitamab+Idelalisib) | Cohort B (Tafasitamab+Venetoclax)
Started | 11 | 13
Completed | 7 | 5
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Cohort A (Tafasitamab+Idelalisib): Tafasitamab in combination with idelalisib
- Cohort B (Tafasitamab+Venetoclax): Tafasitamab in combination with venetoclax
- Total: Total of all reporting groups
Arm/Group | Cohort A (Tafasitamab+Idelalisib) | Cohort B (Tafasitamab+Venetoclax) | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 11
  >=65 years | 8 | 5 | 13
Age, Continuous [Median (Full Range); unit: years] | 69 [51 to 79] | 64 [50 to 77] | 65 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 2 | 4 | 6
  United States | 0 | 6 | 6
  Poland | 5 | 0 | 5
  Italy | 1 | 0 | 1
  United Kingdom | 0 | 2 | 2
  Germany | 3 | 1 | 4
Number of previous systemic treatment lines [Median (Full Range); unit: Lines] | 5 [2 to 9] | 3 [1 to 5] | 4 [1 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events (AEs)
Description: For details please see Section of Adverse Events Overview
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Tafasitamab+Idelalisib) | Cohort B (Tafasitamab+Venetoclax)
Number analyzed (Participants) | 11 | 13
Participants | 11 | 13

2. Secondary Outcome: Best Objective Response Rate (ORR)
Description: ORR = complete response [CR] + partial response [PR]; Local Evaluation
Time Frame: 2 years
Population: Intention-to-treat patient population consists of all enrolled patients. As per study protocol all patients were required to have computed tomography (CT) scans of the neck, chest, abdomen and pelvis to determine tumor response. These were performed at screening, at Day 1 of Cycles 4, 7, 13, and 19, etc. and at end-of-treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A (Tafasitamab+Idelalisib) | Cohort B (Tafasitamab+Venetoclax)
Number analyzed (Participants) | 11 | 13
Percentage of participants
  Intention-to-treat patient population | 90.9 | 76.9
  Pts with tumor response assessment by CT: number analyzed (Participants) | 11 | 10
  Pts with tumor response assessment by CT | 90.9 | 100

3. Secondary Outcome: Number of Participants With Treatment-emergent or Treatment-boosted Anti-MOR00208 Antibody Formation
Description: Number of participants with treatment-emergent or treatment-boosted anti-MOR00208 (anti-tafasitamab) antibody formation
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Tafasitamab+Idelalisib) | Cohort B (Tafasitamab+Venetoclax)
Number analyzed (Participants) | 11 | 13
Participants | 0 | 0

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MOR00208
Description: Mean Cmax of tafasitamab (MOR00208) at Cycle 3 Day 15 (after the weekly dosing of tafasitamab in Cycles 1 to 3 including a loading dose at C1D4)
Time Frame: At Cycle 3 Day 15
Population: All patients with available pharmacokinetic data for Cmax at Cycle 3 Day 15.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A (Tafasitamab+Idelalisib) | Cohort B (Tafasitamab+Venetoclax)
Number analyzed (Participants) | 7 | 9
ng/mL | 278379.9 (118746.34) | 306998.9 (41254.20)

5. Other Pre Specified Outcome: Proportion of Patients With MRD-negativity
Description: Proportion of patients who reached MRD-negativity in peripheral blood
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Tafasitamab+Idelalisib) | Cohort B (Tafasitamab+Venetoclax)
Number analyzed (Participants) | 11 | 13
Participants | 1 | 6

ADVERSE EVENTS:
Time Frame: From the first administration of any study drug to the patient until the 30-day safety follow-up visit as per protocol or until the cut-off date of 09 November 2018 whichever comes first.
Arm/Group | Cohort A (Tafasitamab+Idelalisib) | Cohort B (Tafasitamab+Venetoclax)
All-Cause Mortality (participants affected / at risk) | 2/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 8/11 | 9/13
Other Adverse Events (participants affected / at risk) | 11/11 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Tafasitamab+Idelalisib) (N=11) | Cohort B (Tafasitamab+Venetoclax) (N=13)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Tafasitamab+Idelalisib) (N=11) | Cohort B (Tafasitamab+Venetoclax) (N=13)
Neutropenia (Blood and lymphatic system disorders) | 5 (15) | 6 (21)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Erythema of eyelid (Eye disorders) | 1 (1) | 0 (0)
Holmes-Adie pupil (Eye disorders) | 1 (1) | 0 (0)
Pupils unequal (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Noninfective sialoadenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (8) | 2 (2)
Fatigue (General disorders) | 1 (2) | 3 (3)
General physical health deterioration (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (3) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immunodeficiency (Immune system disorders) | 2 (2) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in liver (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (5) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (3)
Amylase increased (Investigations) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (2) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 4 (4)
Troponin T increased (Investigations) | 0 (0) | 3 (3)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 2 (2)
Coombs test positive (Investigations) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (3) | 2 (4)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small airways disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT02639910/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT02639910/SAP_000.pdf